CLINICAL TRIAL: NCT03787589
Title: A Simple Exercise Program for Patients With End Stage Kidney Disease to Improve Strength and Quality of Life: A Feasibility Study
Brief Title: Exercise in Patients With End Stage Kidney Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 618
Record Dates: First submitted 2018-10-01; First posted 2018-12-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Renal Failure
Keywords: Renal Failure; Hemodialysis; Peritoneal Dialysis; Exercise
MeSH Terms: conditions — Renal Insufficiency; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Participants in this arm will receive standard of care along with the exercise prescription intervention
  Interventions: Behavioral: Exercise Prescription
- Standard of Care (No Intervention): This group will receive standard of care treatment including regular verbal encouragement to exercise (monthly) by dialysis unit staff.

INTERVENTIONS:
Behavioral: Exercise Prescription — Participants in the intervention group will be given an exercise prescription to increase their baseline steps by 1200 and 2000 steps per day at least 3 days a week over the first 3 months. If tolerated and accepted, the participants will increase their step counts by an additional 600 to 1000 steps per day at least 3 days a week for the next 3 months.This will be followed by a 6-month maintenance phase. The research coordinator will instruct the participants on the proper use of the Nordic walking poles which can be used to help participants achieve their prescribed number of steps.
  All participants will be encouraged to wear the pedometer throughout the trial in order to follow the step-count prescription and monitor adherence.
  Arms: Exercise Intervention

SUMMARY:
This study will be conducted over a 3 year time period. This is a trial of an exercise intervention vs. standard of care in patients receiving chronic dialysis. The specific aims will be to determine feasibility of patient recruitment, adherence to the exercise program, and efficacy of the intervention on patient important outcomes.

The exercise intervention will be delivered to randomized participants for 12 months, and consist of the prescribed use of Nordic Walking poles, online resources for exercise in the home, regular use of a pedometer to monitor progress, and regular verbal encouragement to exercise (monthly) by dialysis unit staff. Both groups will receive the same standard of care co-interventions including individualized dialysis prescriptions and health-care interactions according to practices at their centre.

ELIGIBILITY:
Inclusion Criteria:

1. All ambulatory adult patients with end stage kidney disease
2. Treatment with peritoneal dialysis or hemodialysis for greater than six months
3. Able to understand English or French
4. Abuse to use Nordic Walking poles
5. Able and willing to provide informed consent

Exclusion Criteria:

1. Any absolute contraindication to exercise [unstable angina, uncontrolled hypertension (systolic or diastolic blood pressure greater than 180 mmHg (millimeters of mercury) or greater than 110 mmHg, respectively), deemed not suitable for exercise by the treating physician]
2. Baseline step count greater than 8000 steps a day
3. Planned living donor kidney transplant
4. Potential for recovery of renal function
5. Patients who feel unsafe using Nordic walking poles in place of their mobility aid
6. Participation in another interventional trial that may affect the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-15 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | 30 months
  The investigators will assess at each centre the number of participants receiving dialysis, approached for participation, eligible to participate and any reasons for non-participation.
Adherence | 12 months
  Two-week step counts with a pedometer will be monitored monthly in the treatment group, and at baseline, 6 and 12 months in the control group.

SECONDARY OUTCOMES:
Hand Grip Strength | 12 months
  The investigators will measure hand grip strength at baseline, 6, and 12 months using a handgrip dynamometer in the dominant hand or in the non-arteriovenous fistula arm (best of two efforts in kgs)
Quality of Life using Vitality Subscale | 12 months
  Energy will be measured with the Medical Outcomes Study 36 Item Short Form Survey Instrument - Vitality Subscale (Score 0 (lowest) -100 (highest, more energy)
Sleep Quality | 12 months
  Sleep will be measured with the Pittsburgh Sleep Quality Index (Score 0-21; lower scores reflect better sleep).
Hospitalizations | 12 months
  The number of hospitalizations per patient year
Hospital Length of Stay | 12 months
  Average number of days spent in hospital
Change in Living Status | 12 months
  Including full care (admission to a long-term care facility), need for assistance such as housekeeping, meals, bathing
Safety of the Exercise Program | 12 months
  Safety will be measured by monitoring serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Zimmerman, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, manual of operations and consent form will be made available by contacting the corresponding author. De-identified patient data will be available from 12 months to 3 years after manuscript publication to researchers with methodologically sound proposals approved by the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: One year after publication up to 3 years post publication
Access Criteria: researchers with methodologically sound proposals approved by the principal investigator

REFERENCES:
- [Derived] Suri RS, Moist L, Lok C, Clase CM, Harris J, Reid RD, Ramsay T, Zimmerman D. A Simple Exercise Program for Patients With End-Stage Kidney Disease to Improve Strength and Quality of Life: Clinical Research Protocol. Can J Kidney Health Dis. 2023 Oct 26;10:20543581231205160. doi: 10.1177/20543581231205160. eCollection 2023. PMID 37901358